CLINICAL TRIAL: NCT04195386
Title: Efficacy of a Chemically Activated Composite Resin Alkasite in Atypical Caries Lesions of Deciduous Teeth - Randomized Clinical Trial
Brief Title: Efficacy of a Chemically Activated Composite Resin Alkasite in Atypical Caries Lesions of Deciduous Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Principal Investigator, Jose Carlos P Imparato, PhD in Pediatric Dentistry, Faculty Sao Leopoldo Mandic Campinas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLM2990
Record Dates: First submitted 2019-09-30; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Dental Caries in Children
Keywords: Dental caries; Deciduous teeth; Permanent dental restoration
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Compare the survival of restorations performed with chemically activated composite resin alkasite and resin- modified glass ionomer cement.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemically activated Composite resin Alkasite (Experimental): Single placement of composite resin on atypical cavities.
  Interventions: Procedure: Dental Restoration with Chemically activated Composite resin Alkasite
- Resin-Modified Glass ionomer Cement (Active Comparator): Single placement of Resin-Modified Glass ionomer Cement on atypical cavities.
  Interventions: Procedure: Dental Restoration with Resin-Modified Glass ionomer Cement

INTERVENTIONS:
Procedure: Dental Restoration with Chemically activated Composite resin Alkasite — Selective removal of dental caries with manual instruments, under relative isolation, application of universal adhesive system and restoration with chemically activated composite resin Alkasite.
  Arms: Chemically activated Composite resin Alkasite
Procedure: Dental Restoration with Resin-Modified Glass ionomer Cement — Selective removal of dental caries with manual instruments, under relative isolation, application of polyacrylic acid and restoration with resin-modified glass ionomer cement.
  Arms: Resin-Modified Glass ionomer Cement

SUMMARY:
Atypical cavities, which involve more than two surfaces being one of them vestibular or lingual/palatine, are a challenge for restorative dentistry, since the risk of failure of the restorations are related to the number of surfaces involved. Thus, the objective of this project is to conduct a randomized clinical trial in order to evaluate the efficacy and patient-centered outcomes of a chemically-activated alkasite composite resin in atypical lesions of deciduous molars. Deciduous molars of children between 4 and 7 years of age with at least one atypical cavity lesion in deciduous molars will be selected for the ECR. The selected teeth will be randomly divided into two groups: Chemically activated composite resin Alkasite and resin-Modified glass ionomer cement. Clinical and radiographic follow-up of the lesions will be performed for 6 and 12 months. The efficacy of the treatments will be evaluated by the longevity of the restoring procedures and the arrestment of the caries lesions. Patient-centered outcomes will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

• Children will be included who have at least one posterior tooth with atypical caries lesion.

Exclusion Criteria:

* Patients with special needs
* Patients general health conditions that may affect the oral cavity
* Patients non-cooperating in relation to the examination
* Patients with orthodontic apparatus
* The parents/guardians or children not to consent to their participation in the study.
* Teeth with pulp exposure
* Teeth with spontaneous pain
* Teeth with mobility
* Teeth with presence of swelling or fistula close to the tooth
* Teeth with furcation or cervical injury
* Teeth with restorations, sealants or enamel formation defects will be excluded.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Survival of restoration | 12 months after treatment.
  To evaluate the survival of restoration by clinical examination with FDI index.

SECONDARY OUTCOMES:
Caries lesion progression | 12 months after treatment.
  For the evaluation of caries progression, the interproximal radiographic examination will be used to verify an increase of radiolucent image under restoration.
Secondary caries lesion or on the surface adjacent to the restored tooth | 12 months after treatment.
  Presence of caries lesion on the surface adjacent to the restored tooth or on the margins of the restoration by means of visualClinical Examination
Perception of children and parents/guardians | 6 months after treatment.
  To evaluate the satisfaction of the children in relation to the treatment performed. The questionnaire will be used " Child's and parent's questionnaire about teeth appearance".
Operator perception | 6 months after the restoration.
  It will be employed a questionnaire after the completion of the treatment performed. It will also be added a question about the behavior of children during the procedure, which will be categorized as - great behavior, regular or bad.
Parents/Guardians Satisfaction | 6 months after restoration.
  The parents/guardians will be questioned about the satisfaction regarding the treatment performed in the child. The answer will be scored by a likert scale.
Child discomfort | Immediately after the treatment.
  The child will also be questioned as to the discomfort in relation to the treatment performed. For this will be used the scale of faces of Wong-Baker.
Post Operative sensitivity of the child | 7 ° day after the restorative procedure.
  The child will also be questioned about the sensitivity of the restorative procedure. For this, the Wong-Baker face scale will be used.
Oral health-related quality of life | 6 month of restorative treatment.
  The validated Brazilian version of Early Childhood Oral Health Impact Scale (ECOHIS) will be applied to children and should be answered by their parents.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade Sao Leopoldo Mandic, Campinas, São Paulo, Brazil